CLINICAL TRIAL: NCT01432184
Title: Perioperative Interventions to Optimize Cerebral Oxygen Saturation (rSO2) in High-risk Patients Undergoing Cardiac Surgery Should Have a Beneficial Systemic Effect for Enhancing Global Tissue Perfusion and Improve Outcomes.
Brief Title: Feasibility Trial to Maintain Normal Cerebral Oxygen Saturation in High-Risk Cardiac Surgery
Acronym: Tête-à-coeur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Alain Deschamps, PhD, MD, FRCPC,, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICM 08-1009
Record Dates: First submitted 2011-08-26; First posted 2011-09-12 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Cerebral Hypoxia
Keywords: cerebral; hypoxia
MeSH Terms: conditions — Hypoxia, Brain; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): an alarm threshold at a value of 90% of the resting baseline cerebral saturation value (baseline - 10%) will be established. To minimize the probability of patients reaching significant decreases rSO2 values, interventions to improve cerebral oxygenation will be initiated according to the strategies described in the algorithm. The success and failure of these interventions will be noted. As in the Control group, the screen will remain blinded in the ICU and the intensivist will not see the values.
  Interventions: Procedure: strategies to reverse decrease in rSO2
- Control (No Intervention): the cerebral oxymetry screen will be blinded and changes in NIRS values will be unknown to the anesthesiologist. The management of the case will proceed as per normal local practice. The screen will remain blinded in the ICU and the intensivist will not see the values.

INTERVENTIONS:
Procedure: strategies to reverse decrease in rSO2 — an alarm threshold at a value of 90% of the resting baseline cerebral saturation value (baseline - 10%) will be established. To minimize the probability of patients reaching significant decreases rSO2 values, interventions to improve cerebral oxygenation will be initiated according to the strategies described in the algorithm. The success and failure of these interventions will be noted. As in the Control group, the screen will remain blinded in the ICU and the intensivist will not see the values.
  Other Names: Cerebral Oxymetry decrease
  Arms: Intervention

SUMMARY:
Using the brain and the heart as index organs, perioperative interventions to optimize cerebral oxygen saturation and cardiac contractility in high-risk patients undergoing cardiac surgery should have a beneficial systemic effect for enhancing global tissue perfusion and improve outcomes.

DETAILED DESCRIPTION:
The proportion of high-risk patients requiring cardiac surgery and of high-risk cardiac surgeries is increasing. These populations of patients are at increased risk of perioperative morbidity and mortality. Transesophageal echocardiography (TEE) evaluation in cardiac surgery has been shown to impact on the perioperative management of patients and to improve outcomes. Near infrared-reflectance spectroscopy (NIRS) is a technique that has been employed since the mid-1970's and that can be used as a non-invasive and continuous monitor of the balance between cerebral oxygen delivery and consumption. Two recent randomized trials have shown an association between correction of cerebral desaturation and shorter recovery room and hospital stay in non-cardiac surgery, and with a decrease in major organ dysfunction and in intensive care length of stay after coronary artery bypass. By combining NIRS and TEE in high-risk patients, optimal tissue perfusion could be achieved and perioperative morbidity and mortality could be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Patients with EUROSCORES ≥ 10.
* Planned complex surgery including more than one procedure, or redo procedures.
* Patient able to read and understand the consent form.
* Patients ≥ 18 years of age.

Exclusion Criteria:

* High risk patients undergoing of off pump coronary artery bypass.
* Emergency surgeries less than 6 hours from diagnosis.
* Patient unable to read and understand the consent form.
* Patients with and IABP or a ventricular assist device
* Planned circulatory arrest
* Planned surgery of the descending aorta.
* Patients with acute endocarditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-07; Primary Completion 2011-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Success rate of reversing decreases in cerebral oxygen saturation below 10% of baseline values to values within 10% of baseline in the INTERVENTION group. | Up to 12 hours
  Consensus on the appropriate strategies to prevent and reverse cerebral oxygen desaturations remains controversial. In a recent study by Slater and al.12, randomization into an intervention group failed because anesthesiologists were unable to follow the protocol aimed at strategies to reverse decreases in rSO2. A group from the Montreal Heart Institute has developed a physiologically oriented algorithm to help with the task of reversing decreases in rSO2. The goal of the present study is therefore to confirm that this approach can be used with success by most institutions.

SECONDARY OUTCOMES:
First 30 days post-operative outcomes | 30 days
  * readmission to hospital within 30 days
  * death
ICU data | Up to 48 hours
  * ICU admission and discharge times
  * tracheal extubation time in hours
First 24 hours complications | 24 hours
  * clinical stroke manifested as focal neurological deficit persisting 24hr and confirmed by brain computed tomography imaging
  * prolonged ventilation defined as extubation at > 24 h postoperatively
  * new, persistent Q-wave myocardial infarction
Post-operative complications | Up to 7 days
  * renal failure as defined by the RIFLE criteria
  * reoperation for any cause
  * arrhythmia requiring treatment
  * Hospital length of stay
  * wound infection requiring specific antibiotic coverage

CONTACTS AND LOCATIONS:
Overall Officials: Alain Deschamps, MD, FRCPC, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Taillefer MC, Denault AY. Cerebral near-infrared spectroscopy in adult heart surgery: systematic review of its clinical efficacy. Can J Anaesth. 2005 Jan;52(1):79-87. doi: 10.1007/BF03018586. PMID 15625262
- [Background] Kurth CD, Steven JL, Montenegro LM, Watzman HM, Gaynor JW, Spray TL, Nicolson SC. Cerebral oxygen saturation before congenital heart surgery. Ann Thorac Surg. 2001 Jul;72(1):187-92. doi: 10.1016/s0003-4975(01)02632-7. PMID 11465176
- [Background] Hadolt I, Litscher G. Noninvasive assessment of cerebral oxygenation during high altitude trekking in the Nepal Himalayas (2850-5600 m). Neurol Res. 2003 Mar;25(2):183-8. doi: 10.1179/016164103101201175. PMID 12635520
- [Background] Casati A, Fanelli G, Pietropaoli P, Proietti R, Tufano R, Danelli G, Fierro G, De Cosmo G, Servillo G; Collaborative Italian Study Group on Anesthesia in Elderly Patients. Continuous monitoring of cerebral oxygen saturation in elderly patients undergoing major abdominal surgery minimizes brain exposure to potential hypoxia. Anesth Analg. 2005 Sep;101(3):740-747. doi: 10.1213/01.ane.0000166974.96219.cd. PMID 16115985
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Denault A, Deschamps A, Murkin JM. A proposed algorithm for the intraoperative use of cerebral near-infrared spectroscopy. Semin Cardiothorac Vasc Anesth. 2007 Dec;11(4):274-81. doi: 10.1177/1089253207311685. PMID 18270192
- [Background] Jobsis FF. Non-invasive, infra-red monitoring of cerebral O2 sufficiency, bloodvolume, HbO2-Hb shifts and bloodflow. Acta Neurol Scand Suppl. 1977;64:452-3. No abstract available. PMID 268870
- [Background] Edmonds HL Jr, Ganzel BL, Austin EH 3rd. Cerebral oximetry for cardiac and vascular surgery. Semin Cardiothorac Vasc Anesth. 2004 Jun;8(2):147-66. doi: 10.1177/108925320400800208. PMID 15248000
- [Background] Sokol DK, Markand ON, Daly EC, Luerssen TG, Malkoff MD. Near infrared spectroscopy (NIRS) distinguishes seizure types. Seizure. 2000 Jul;9(5):323-7. doi: 10.1053/seiz.2000.0406. PMID 10933986
- [Background] Shojima M, Watanabe E, Mayanagi Y. Cerebral blood oxygenation after cerebrospinal fluid removal in hydrocephalus measured by near infrared spectroscopy. Surg Neurol. 2004 Oct;62(4):312-8; discussion 318. doi: 10.1016/j.surneu.2003.09.035. PMID 15451273
- [Background] Gracias VH, Guillamondegui OD, Stiefel MF, Wilensky EM, Bloom S, Gupta R, Pryor JP, Reilly PM, Leroux PD, Schwab CW. Cerebral cortical oxygenation: a pilot study. J Trauma. 2004 Mar;56(3):469-72; discussion 472-4. doi: 10.1097/01.ta.0000114274.95423.c0. PMID 15128115
- [Background] Vernieri F, Tibuzzi F, Pasqualetti P, Rosato N, Passarelli F, Rossini PM, Silvestrini M. Transcranial Doppler and near-infrared spectroscopy can evaluate the hemodynamic effect of carotid artery occlusion. Stroke. 2004 Jan;35(1):64-70. doi: 10.1161/01.STR.0000106486.26626.E2. Epub 2003 Dec 18. PMID 14684777
- [Background] Yao FS, Tseng CC, Ho CY, Levin SK, Illner P. Cerebral oxygen desaturation is associated with early postoperative neuropsychological dysfunction in patients undergoing cardiac surgery. J Cardiothorac Vasc Anesth. 2004 Oct;18(5):552-8. doi: 10.1053/j.jvca.2004.07.007. PMID 15578464
- [Background] Slater JP, Guarino T, Stack J, Vinod K, Bustami RT, Brown JM 3rd, Rodriguez AL, Magovern CJ, Zaubler T, Freundlich K, Parr GV. Cerebral oxygen desaturation predicts cognitive decline and longer hospital stay after cardiac surgery. Ann Thorac Surg. 2009 Jan;87(1):36-44; discussion 44-5. doi: 10.1016/j.athoracsur.2008.08.070. PMID 19101265
- [Background] de Tournay-Jette E, Dupuis G, Bherer L, Deschamps A, Cartier R, Denault A. The relationship between cerebral oxygen saturation changes and postoperative cognitive dysfunction in elderly patients after coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2011 Feb;25(1):95-104. doi: 10.1053/j.jvca.2010.03.019. Epub 2010 Jul 22. PMID 20650659
- [Background] Deschamps A, Rochon A, Lebon J-S, Ayoub C, Qizilbash B, Couture P, Cogan J, Toledano K, Bélisle S, Hemmings G, Taillefer J, Blain R, Denault A: Decreases in Cerebal Oxygen Saturation: an algorithmic approach. Canadian Anaesthetists' Society Journal 2009; Abstract: #613224
- [Background] Fergusson DA, Hebert PC, Mazer CD, Fremes S, MacAdams C, Murkin JM, Teoh K, Duke PC, Arellano R, Blajchman MA, Bussieres JS, Cote D, Karski J, Martineau R, Robblee JA, Rodger M, Wells G, Clinch J, Pretorius R; BART Investigators. A comparison of aprotinin and lysine analogues in high-risk cardiac surgery. N Engl J Med. 2008 May 29;358(22):2319-31. doi: 10.1056/NEJMoa0802395. Epub 2008 May 14. PMID 18480196